CLINICAL TRIAL: NCT00459888
Title: CLIMB Prospective Multicenter Registry Evaluating the Use of the PolarCath Peripheral Dilatation System (Boston Scientific) in the Treatment of Infrapopliteal Lesions in Patients With Critical Limb Ischemia (Rutherford 4 and 5).
Brief Title: Cryoplasty CLIMB-registry
Acronym: CLIMB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Flanders Medical Research Program (FMRP)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-001
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Occlusive Disease
Keywords: CLI; Critical Limb Ischemia; Infrapopliteal; Cryoplasty
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PolarCath Peripheral Dilatation System (Boston Scientific)

SUMMARY:
In 5 Belgian hospitals, the data of 100 CLI-patients receiving the cryoplasty technique to treat their infrapopliteal arterial lesions will be collected. The treatment occurs strictly according the "Instructions For Use" of the CE-approved device (PolarCath Peripheral Dilatation System, Boston Scientific) and only data are collected that have been made available conform the Standard the Standards of Care for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic CLI male or female patients with at least 1 atherosclerotic diseased infrapopliteal artery. If patients present with more than 1 diseased vessel, only the vessel with the best distal run-off providing the foot with blood, will be assessed following treatment with the PolarCath Peripheral Dilatation System (Boston Scientific) and analysed for registry purposes.

Patients will be considered eligible for inclusion into the registry if satisfying the product DFU specifications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Clinical patency | 12 months

SECONDARY OUTCOMES:
Technical success | procedure
angiographic outcomes for the subgroup of patients in which made available. | 12 months
Primary patency rate | 12 months
Limb-salvage rate | 12 months
Serious adverse events | 12 months
Clinical success (improvement of Rutherford classification) | 12 months
Health Economics assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint-Blasius, Dendermonde, Belgium; Frank Vermassen, MD, Principal Investigator — University Hospital Ghent, Belgium
Locations (4):
- Belgium (4):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - ZOL Campus Sint-Jan, Genk
  - University Hospital, Ghent

REFERENCES:
- [Derived] Bosiers M, Deloose K, Vermassen F, Schroe H, Lauwers G, Lansinck W, Peeters P. The use of the cryoplasty technique in the treatment of infrapopliteal lesions for Critical Limb Ischemia patients in a routine hospital setting: one-year outcome of the Cryoplasty CLIMB Registry. J Cardiovasc Surg (Torino). 2010 Apr;51(2):193-202. PMID 20354489